CLINICAL TRIAL: NCT05903612
Title: A Prescreening Study to Diagnose Allergic Bronchopulmonary Aspergillosis in Selected Patients With Asthma
Brief Title: Allergic Bronchopulmonary Aspergillosis Prescreening Study
Status: Withdrawn | Type: Observational
Why Stopped: Reasons unrelated to safety issues
Sponsor: Community Pharmacology Services Ltd (Other)
Collaborators: Pulmatrix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 601-0023
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Allergic Bronchopulmonary Aspergillosis; Asthma; ABPA
Keywords: ABPA; Allergic Bronchopulmonary Aspergillosis; Asthma
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prescreening study is being conducted to diagnose ABPA in selected patients with asthma and to increase the potential number of eligible participants for the ongoing Study 601-0018 of PUR1900 in subjects with ABPA. See: NCT05667662.

Additionally, this prescreening study may provide information that could assist the conduct of future studies conducted by Pulmatrix.

DETAILED DESCRIPTION:
See NCT05667662 for a detailed description fo the main ABPA study. This prescreening study is designed to diagnose ABPA in patients with asthma to potentially increase the number of eligible participants for the ongoing NCT05667662 study. This diagnosis will be confirmed through chest x-rays and a blood sample.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent before the performance of any study-specific procedures at the in-clinic visit.
2. Is a male or female ≥18 years old.
3. Has a BMI of ≥18.0 and <40.0 kg/m2 at the in-clinic visit.
4. Meets the following criteria:

   1. Has a diagnosis of asthma.
   2. At least 1 exacerbation requiring a systemic glucocorticosteroid(s) or hospital admission in the last 10 months.
   3. For patients on a biologic agent, at least one exacerbation requiring a systemic glucocorticosteroid(s) or hospital admission must have occurred at least 3 months after the initiation of the biologic agent.
5. Is willing and able to comply with all study procedures

Exclusion Criteria:

1. Has used omalizumab (Xolair®) in the 11 months prior to screening or plans to use omalizumab during the study.
2. Has a current diagnosis of any chronic airway disease other than asthma, ABPA, or bronchiectasis believed to be related to ABPA, such as chronic obstructive pulmonary disease, pulmonary fibrosis, CF, or Churg-Strauss syndrome.
3. Currently requiring medications that are sensitive substrates for CYP3A4-mediated metabolism or medications that are contraindicated during and 2 weeks after treatment with oral formulations of itraconazole without the possibility of washout (See Appendix 4).
4. Smoking marijuana or tobacco, the use of e-cigarettes, vaping, or any other smoking is prohibited during the study.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled at study sites in North America, Europe, and the Asia-Pacific region participating in Study 601-0018. Only patients who meet all eligibility criteria will be enrolled in the prescreening study and have blood samples drawn for laboratory testing at the in-clinic visit.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Patients Diagnosed | 6 weeks
  Number of patients with known asthma and diagnosis of ABPA
Patients Invited | 6 weeks
  Number of patients invited to participate in Study 601-0018

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Wasilewski, MD, Study Director — Pulmatrix Inc.
Locations (1):
- CPS Research, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No